CLINICAL TRIAL: NCT03911960
Title: Acceptance and Commitment Therapy for Tobacco Cessation Initiated in a Psychiatric Partial Hospital
Brief Title: Acceptance and Commitment Therapy for Tobacco Cessation Among Psychiatric Partial Hospital Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03DA043596-01A1 (NIH)
Record Dates: First submitted 2019-03-26; First posted 2019-04-11 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2019-01

CONDITIONS: Tobacco Smoking; Psychiatric Disorder; Psychiatric Hospitalization
Keywords: tobacco smoking; psychiatric disorder; psychiatric hospitalization; acceptance and commitment therapy
MeSH Terms: conditions — Tobacco Smoking; Mental Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): 2 in person and 5 telephone sessions of Acceptance and Commitment Therapy for tobacco cessation plus up to 8 weeks of nicotine patch.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Enhanced Usual Care (Active Comparator): 2 in-person sessions of tobacco cessation counseling, electronic referral to state quitline, up to 8 weeks of nicotine patch
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — 2 in person and 5 telephone sessions of acceptance and commitment therapy for tobacco cessation plus up to 8 weeks of nicotine patch
  Arms: Acceptance and Commitment Therapy
Behavioral: Enhanced Usual Care — 2 in person sessions of tobacco cessation counseling, up to 8 weeks of nicotine patch, referral to state quitline.
  Arms: Enhanced Usual Care

SUMMARY:
People with serious mental illness are three times more likely to smoke cigarettes than people without mental illness. People with mental illness are less likely to be successful in quitting smoking than those without mental illness. Therefore, the healthcare community needs to find ways to get people with mental illness treatment to help them stop smoking. This study explores whether a treatment, called acceptance and commitment therapy, which is an affective therapy for serious mental illness, can help patients with serious mental illness stop smoking. In particular, the investigators test whether patients will be interested in receiving acceptance and commitment therapy for smoking cessation in a psychiatric partial hospital (also known as a day treatment program), whether they are able to complete the treatment, and whether it will help them stop smoking compared to usual care. To test these research questions, 40 patients in the Rhode Island Hospital's psychiatric partial hospital will be recruited. Half of the patients will receive acceptance and commitment therapy to help them stop smoking (2 in person sessions, 5 telephone sessions) and half will receive usual care (2 in person sessions, electronic referral to the Rhode Island tobacco quit line). All participants will be offered the nicotine patch. All participants will complete a baseline survey and a follow-up visit at the end of treatment to measure whether they stopped smoking and whether they liked the treatment. The study will also measure how many participants completed the treatment sessions. If successful, this treatment model could be a way to get more patients with mental illness into treatment.

DETAILED DESCRIPTION:
BACKGROUND: There is a significant disparity in tobacco use in that smokers with mental illness smoke at twice the rate of the general population, use more tobacco per day and are disproportionately affected by smoking-related disease. Few models exist for treating tobacco use in individuals with mental illness. Acceptance and Commitment Therapy (ACT) is a treatment strategy that helps individuals accept discomfort while making value-guided change. It has been used successfully to treat psychiatric symptoms in people with serious mental illness (SMI) and is well-suited to treat smoking in people with SMI. Psychiatric partial hospitalization programs provide an opportunity to intervene on tobacco use in people with SMI. OBJECTIVE: This study tests the feasibility of offering an ACT-based smoking cessation treatment initiated in a psychiatric partial hospital program and continuing post-discharge. AIMS: The study has 3 aims: (1) To assess the feasibility, acceptability, and safety of an ACT-based, partial hospital initiated, counseling intervention for smoking cessation. (2) To collect preliminary evidence of the efficacy (i.e., effect size estimates) of ACT-based counseling initiated in the partial hospital compared to usual care. (3) To explore of the effect of treatment condition (ACT vs. Usual Care) on ACT treatment targets. DESIGN: This study is a randomized design (n=40), where patients in an ACT-based psychiatric partial hospital will be offered up to 8 weeks of the nicotine patch and randomly assigned to either ACT care (n=20; two in-person ACT-based counseling sessions + 5 ACT-based telephone counseling sessions) or to Enhanced Usual Care (n=20; two in person medication management counseling sessions + referral to the state quit line). Outcomes assessed at end of treatment include: feasibility (percent of eligible patients who enroll, percent of patients completing treatment), acceptability (patient satisfaction ratings), safety (hospital readmissions, symptom exacerbation), efficacy (CO confirmed 7 day point prevalence abstinence at end of treatment) and ACT treatment targets (tolerance of discomfort, mindfulness and acceptance). SIGNIFICANCE: This study tests a treatment model for smokers with SMI, a group with particularly refractory smoking behavior. If successful, this model could be implemented broadly in psychiatric day treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and female
* psychiatry partial hospital patients
* current daily smokers

  -≥ age 18
* have regular telephone access
* able to read and write English

Exclusion Criteria:

-current use of tobacco cessation treatment (bupropion prescribed for a psychiatric indication will be permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Japuntich, Ph.D., Principal Investigator — Hennepin Healthcare Research Institute; Ernestine Jennings, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Only the Principal Investigator will give permission for the release of aggregated study data. No identifiable data will be released. Participants in the proposed research will be informed, during consent, that completely de-identified data (i.e., data that has been cleaned of all 18 types of HIPAA identifiers) will be available to other qualified researchers. Within 18 months of study completion, we will make datasets available to interested investigators who submit a written request to the PI. The only contingency on the use of the data will be that ethical guidelines be followed (e.g., only individuals who have completed a research ethics training course will have access to the data, the data will be stored securely). The NIH will be notified of transmissions of the data to interested investigators.
Supporting Information: Study Protocol, ICF
Time Frame: within 18 months of study completion
Access Criteria: ethical guidelines for The Miriam Hospital will be followed (the investigator will have completed a research ethics training course and the data will be stored securely)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 participants consented to the study and were randomized but completed none of the study procedures (did not complete the baseline questionnaire, any of the counseling sessions, or the follow-up visit).
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Started | 9 | 5
Completed | 4 | 2
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.33 (17.30) | 34.00 (12.39) | 38.71 (15.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment: Proportion of Smokers Seen During the Partial Hospital Visit Who Enroll in the Study
Description: proportion of smokers seen during the partial hospital visit who enroll in the study
Time Frame: Through study completion, approximately 5 months.
Population: This analysis calculates the number of smokers screened in the partial hospitalization program who participated in the trial
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: This outcome assesses interest in the trial prior to randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 66
Participants | 17

2. Primary Outcome: Percentage of Counseling Sessions Completed
Description: number of scheduled counseling sessions completed
Time Frame: through study completion, an average of 7 weeks.
Measure: Number; unit: percentage of sessions completed
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 9 | 5
percentage of sessions completed | 48 | 80

3. Primary Outcome: Client Satisfaction Questionnaire
Description: The Client satisfaction Questionnaire, measures acceptability of the intervention to patients, minimum value=8, maximum value=32, higher scores indicate higher satisfaction (higher scores mean better outcome)
Time Frame: at study completion, an average of 7 weeks post-enrollment
Population: participants who completed the follow-up questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 4 | 2
units on a scale | 27.00 (6.63) | 27.5 (0.71)

4. Primary Outcome: Number of Participants Who Are Rehospitalized for Psychiatric Reasons
Description: This is a simple count based on follow-up survey data of the number of participants who reported being hospitalized for a psychiatric reason following enrollment in the study.
Time Frame: At study completion, an average of 7 weeks post enrollment
Population: participants who completed the follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Who Are Abstinent From Tobacco
Description: a simple count of those who have both a carbon monoxide value consistent with abstinence and self-reported abstinence. Expired carbon monoxide value of less than 6 parts per million was considered abstinent.
Time Frame: at study completion, an average of 7 weeks post enrollment
Population: all participants who started the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 9 | 5
Participants | 1 | 0

6. Secondary Outcome: Kessler 6
Description: Kessler 6, global distress measure, minimum value=0, maximum value=24, higher scores = greater distress (worse outcome), this study measures the change in global distress between enrollment and study completion. The change in global distress score minimum value=-24, maximum value=24 (lower scores indicate a better outcome: a reduction in distress)
Time Frame: Change between baseline and study completion, 7 weeks post-enrollment
Population: participants who completed follow-up assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 4 | 2
units on a scale | -4.25 (7.59) | -5.0 (7.07)

7. Other Pre Specified Outcome: Avoidance Inflexibility Scale
Description: The avoidance inflexibility scale is a 13-item self-report assessment in which respondents to consider how they respond to difficult thoughts that encourage smoking (e.g., "I need a cigarette", "I wish I could have a cigarette now!"), different feelings that encourage smoking (e.g., stress, fatigue, boredom, enjoyment, satisfaction, etc.), and bodily sensations that encourage smoking (e.g., "physical cravings or withdrawal symptoms").The Avoidance Inflexibility Scale measures smoking-related experiential avoidance, minimum score= 13, maximum score=65, higher score indicate more avoidance (worse outcome), the study outcome is the change between avoidance measured at baseline, and at study completion, 7 weeks post-enrollment. Minimum score=-52, maximum score=52 lower scores = better outcome.
Time Frame: Change between baseline and study completion, 7 weeks post-enrollment
Population: people who completed follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 4 | 2
units on a scale | -9.25 (15.69) | 6.5 (6.36)

8. Other Pre Specified Outcome: Commitment to Quitting Scale
Description: Commitment to Quitting Scale, range 8-40, higher scores indicate greater commitment, commitment will be measured as the change between baseline and study completion, 7 weeks post enrollment.
Time Frame: Change between baseline and study completion, 7 weeks post-enrollment
Population: participants who completed the follow-up survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
Number analyzed (Participants) | 4 | 2
units on a scale | 4.25 (7.63) | 4.5 (4.95)

ADVERSE EVENTS:
Time Frame: 5 weeks (from enrollment to follow-up)
Arm/Group | Acceptance and Commitment Therapy | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03911960/ICF_001.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03911960/SAP_002.pdf
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03911960/Prot_003.pdf